CLINICAL TRIAL: NCT02569996
Title: A Multicenter, Phase III, Open-label Study Evaluating the Benefit of a Long-term Effect of MabThera (Rituximab) Maintenance Therapy in Patients With Advanced Follicular Lymphoma After Induction of Response (CR[u] or PR) With MabThera (Rituximab) Containing First-line Regimen
Brief Title: A Study of Long-Term Rituximab (MabThera) Maintenance Therapy in Participants With Advanced Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18167
Record Dates: First submitted 2015-09-23; First posted 2015-10-07 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

ARMS (1):
- Rituximab (Experimental): Participants will receive rituximab 375 milligrams per meter square (mg/m^2) every 8 weeks for 24 months or until progression, relapse, death, or institution of a new anti-lymphoma treatment.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered at 375 mg/m^2 every 8 weeks for 24 months or until progression, relapse, death, or institution of a new anti-lymphoma treatment.
  Other Names: MabThera/Rituxan

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of long-term maintenance therapy with rituximab in participants with advanced follicular lymphoma who have had a positive response to first-line treatment with a rituximab-containing regimen. The anticipated time on study treatment is 2 years, and the target sample size is 124 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than (>) 18 years of age
* Histologically confirmed follicular lymphoma Grade 1, 2, or 3a with lymph node biopsy within 4 months of induction treatment
* No previous anti-lymphoma treatment before induction chemotherapy (first-line-treated participants only are eligible)
* Verified complete or partial remission after first-line induction therapy including rituximab

Exclusion Criteria:

* Grade 3b follicular lymphoma
* Transformation to high-grade lymphoma (except to Grade 3a) of previously existing follicular lymphoma
* Presence of central nervous system lymphoma
* Acquired immunodeficiency syndrome-related lymphoma
* Other primary malignancy (other than squamous cell cancer of the skin or in situ cancer of the cervix) for which the participant has not been disease-free for greater than or equal to (>=) 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2005-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (16):
- Hungary (16):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Veszprém
  - Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 08 July 2005 to 12 Aug 2013 at 15 sites in Hungary.
Pre-assignment Details: A total number of 124 patients were recruited. Of these, 83 patients completed the maintenance therapy with rituximab (MabThera) and entered the 3-year follow-up phase. Of these, 69 patients completed the follow-up phase.
Groups:
- Rituximab: Participants received rituximab 375 milligrams per meter square (mg/m^2) every 8 weeks for 24 months
Period: Overall Study
Arm/Group | Rituximab
Started | 124
Completed | 69
Not Completed | 55
Not completed — Adverse Event | 6
Not completed — Physician Decision | 3
Not completed — Progression of the disease | 18
Not completed — New anti-lymphoma treatment | 1
Not completed — Non-compliance | 9
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 5
Not completed — Complete remission | 7
Not completed — Unknown reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 102
  >=65 years | 22
Age, Continuous [Median (Full Range); unit: years] | 53 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival (EFS) was defined as the time from baseline (Week 0) to the time to progression, relapse, death from any cause, or institution of a new treatment, whichever occurs first. Mean EFS was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval. ITT population (patients who received at least one maintenance MabThera infusion) was used for this analysis.
Time Frame: From randomization to the time to progression, relapse, death from any cause, or institution of a new treatment, whichever occurs first, assessed up to 5 years
Population: ITT population: All participants who received at least one maintenance rituximab infusion were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 124
months | 53.944 [50.242 to 57.647]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, requires intervention to prevent permanent impairment or damage, or results in death
Time Frame: Up to 27 months
Population: Safety population: All participants who received at least one dose of study medication and had safety data after the first dose of study drug.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 124
participants
  SAEs | 14
  Non serious AEs | 32

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival, defined as the time between baseline (Week 0) and the date of death irrespective of the cause of death. Mean OS was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval. ITT population was used for this analysis.
Time Frame: From randomization until death, assessed up to 5 years
Population: ITT population: All participants who received at least one maintenance rituximab infusion were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 124
months | 72.959 [70.303 to 75.616]

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) defined as time from baseline to disease progression or relapse, death from the follicular lymphoma or institution of a new regimen because of the follicular lymphoma. Mean TTP was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval. ITT population was used for this analysis.
Time Frame: From baseline (Week 0) to disease progression, relapse, death from the follicular lymphoma or institution of a new regimen, whichever occurs first, assessed up to 5 years
Population: ITT population: All participants who received at least one maintenance rituximab infusion were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 124
months | 56.024 [52.532 to 59.516]

5. Secondary Outcome: Time to Next Anti-lymphoma Treatment (TTNLT)
Description: Time to next anti-lymphoma treatment (TTNLT) defined as time from baseline to institution of a new antilymphoma regimen (including chemo-, radio- or immunotherapies). Mean TTNLT was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval.
Time Frame: From baseline (Week 0) to institution of a new antilymphoma regimen, assessed up to 5 years
Population: ITT population: All participants who received at least one maintenance rituximab infusion were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 124
months | 59.236 [56.318 to 62.153]

6. Secondary Outcome: Duration of Response (DR)
Description: Duration of Response (DR) defined as time from first documented response to induction treatment to relapse or progression or death from the follicular lymphoma. Mean DR was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval.
Time Frame: From first documented response to induction treatment to relapse or progression or death, assessed up to 5 years
Population: ITT population: All participants who received at least one maintenance rituximab infusion were included in the analysis. Subset of the ITT population was used since not the entire ITT population provided appropriate data for analysis
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 122
months | 63.159 [59.29 to 67.029]

7. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease free survival (DFS) being defined as time from first documented complete response to induction treatment to relapse or progression or death from the follicular lymphoma. Mean DFS was estimated by the Kaplan-Meier estimation and provided with their 95% confidence interval.
Time Frame: From first documented complete response to induction treatment to relapse or progression or death, whichever occurs first, assessed up to 5 years
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 77
months | 66.737 [63.808 to 69.666]

ADVERSE EVENTS:
Time Frame: Up to 27 months
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 14/124
Other Adverse Events (participants affected / at risk) | 3/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=124)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Acute hepatitis B (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Strongyloidiasis (Infections and infestations) | 1
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=124)
Diabetes mellitus (Endocrine disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No